CLINICAL TRIAL: NCT03133884
Title: Acupuncture for Patients With Chronic Tension-type Headache : a Randomized Controlled Trial
Brief Title: Acupuncture for Patients With Chronic Tension-type Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016HH0007
Record Dates: First submitted 2017-03-22; First posted 2017-04-28 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Chronic Tension-Type Headache
Keywords: chronic tension-type headache; acupuncture; Deqi
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): The needles will be inserted into the acupoints and the depths will be adjusted to the standard permissible layers, then even reinforcing-reducing technique will be performed on the needles until achieving deqi sensation.The needles will be retained for 30 minutes in each session and manipulated twice every 10 minutes with intermittent stimulation. Each manipulation will last for 20 seconds.
  Interventions: Other: acupuncture
- Superficial acupuncture (Other): The selected acupoints will be punctured superficially by the depth of 1-3 mm, and the needles will be retained for 30 minutes without any manipulation.
  Interventions: Other: superficial acupuncture

INTERVENTIONS:
Other: acupuncture — The needles will be inserted into the acupoints and the depths will be adjusted to the standard permissible layers, then even reinforcing-reducing technique will be performed on the needles until achieving deqi sensation.The needles will be retained for 30 minutes in each session and manipulated twice every 10 minutes with intermittent stimulation. Each manipulation will last for 30 seconds.
  Arms: Acupuncture
Other: superficial acupuncture — The selected acupoints will be punctured superficially by the depth of 1-3 mm, and the needles will be retained for 30 minutes without any manipulation.
  Arms: Superficial acupuncture

SUMMARY:
Two hundred and eighteen patients with chronic tension-type headache(CTTH) will be randomly assigned to an experimental group (acupuncture) and a control group (superficial acupuncture) in a 1:1 ratio. Participants in both groups will receive 20 sessions of acupuncture over 8 weeks, and the same acupoints will be selected in acupuncture treatments.The study cycle will last 36 weeks, including a 4-week baseline period, a 8-week treatment period and a 24-week follow-up period. And the primary outcome will be measured at the end of 16th week. While, the secondary outcomes will be measured at the baseline, the 4th, 8th,12th,16th,20th,24th,28th and 32nd week after randomization.After each treatment, participants will finish the Massachusetts General Hospital (MGH) Acupuncture Sensation Scale (MASS) to evaluate deqi sensations.

DETAILED DESCRIPTION:
This is a clinical randomized controlled trial (RCT). According to the pervious study, 218 patients, who meet the diagnostic criteria of CTTH in the international classification of headache disorders, 3rd edition (beta version) (ICHD-III beta), will be recruited in this study. And these participants will be randomly assigned to 2groups with acupuncture treatment or superficial acupuncture treatment through central randomization in a 1:1 ratio.

The total observation period will last 36 weeks, including a 4-week baseline period, a 8-week treatment period and a 24-week follow-up period. The central randomization will be performed after the baseline period, and participants will receive 20 sessions of intervention over 8 weeks ( 3 sessions per week in the first 4 weeks and 2 sessions per week in the following 4 weeks).

The same acupoints, named Fengchi (GB20), Taiyang (EX-HN5), Baihui (DU20), Hegu (LI4) and Taichong (LR3) on both sides, will be punctured by filiform needles. However, manipulation methods will be different. In acupuncture group, the needles will be inserted into the acupoints, of which the depths will be adjusted to the standard permissible layers.Then even reinforcing-reducing technique will be performed on the needles until achieving deqi sensation.The needles will be retained for 30 minutes in each session and manipulated twice every 10 minutes with intermittent stimulation. Each manipulation will last for 30 seconds. While, in superficial group, the selected acupoints will be punctured superficially by the depth of 1-3 mm, and the needles will be retained for 30 minutes without any manipulation.

Within 5 minutes after withdrawing needles of each session, participants in three acupuncture groups will finish the Massachusetts General Hospital (MGH) Acupuncture Sensation Scale (MASS).

Most of the curative outcomes will be collected from the headache dairy which is filled by participants. And the primary outcome will be measured at the end of 16th week. While, the secondary outcomes will be measured at the baseline, the 4th, 8th,12th,16th,20th,24th,28th and 32nd week after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting the diagnostic criteria of CTTH in the international classification of headache disorders, 3rd edition (beta version) (ICHD-III beta);
2. Aged 18-65 years;
3. Having the ability of understanding and completing the headache dairy;
4. Volunteering to this study and able to provide written informed consent.

Exclusion Criteria:

1. Not suffering tension-type headache during the pervious 3 months;
2. Taking any prophylactic headache medication during the previous one month;
3. Headache due to organic disorders (e.g. subarachnoid hemorrhage, cerebral hemorrhage, cerebral embolism, cerebral thrombosis, vascular malformation, arthritis, hypertension, arteriosclerosis);
4. Having serious diseases of the heart, liver, kidney or other organs;
5. In pregnancy or lactation, or planning to be pregnant in 6 months;
6. In unconsciousness, or having psychosis;
7. Having bleeding disorders or getting infectious;
8. Unwilling to take parts in this study or with low compliance;
9. Addicted to smoking, alcohol or drugs;
10. Taking parts in other clinical studies at the same time.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Responder rate | 16 weeks after randomization
  The responder rate is defined as >50% reduction in the number of headache days per four week

SECONDARY OUTCOMES:
The number of days with headache | at baseline before randomization, 4, 8, 12, 16, 20, 24, 28 and 32 weeks after randomization
The mean pain intensity of tension-type headache during 4 weeks | at baseline before randomization, 4, 8, 12, 16, 20, 24, 28 and 32 weeks after randomization
  Using a visual analogue scale from 0-10, 0 defined as no pain and 10 defined as an unbearable pain.
The rate of medication intake during 4 weeks | at baseline before randomization, 4, 8, 12, 16, 20, 24, 28 and 32 weeks after randomization
Evaluation of quality of life | at baseline before randomization, 4, 8, 12, 16, 20, 24, 28 and 32 weeks after randomization
  The 36-item short from health survey (SF-36)
Evaluation of anxiety state | at baseline before randomization, 4, 8, 12, 16, 20, 24, 28 and 32 weeks after randomization
  Hamilton anxiety scale (HAMA)
Evaluation of depression state | at baseline before randomization, 4, 8, 12, 16, 20, 24, 28 and 32 weeks after randomization
  Hamilton depression scale (HAMD)
Evaluation of needling sensation | Within 5 minutes after withdrawing needles of each acupuncture session
  the Massachusetts General Hospital (MGH) Acupuncture Sensation Scale (MASS)

CONTACTS AND LOCATIONS:
Overall Officials: Ying Li, PhD, Study Chair — Chengdu University of Traditional Chinese Medicine
Locations (1):
- Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zheng H, Gao T, Zheng QH, Lu LY, Hou TH, Zhang SS, Zhou SY, Hao XY, Wang L, Zhao L, Liang FR, Li Y. Acupuncture for Patients With Chronic Tension-Type Headache: A Randomized Controlled Trial. Neurology. 2022 Oct 3;99(14):e1560-e1569. doi: 10.1212/WNL.0000000000200670. PMID 35732505
- [Derived] Lu L, Zheng H, Zheng Q, Hao X, Zhou S, Zhang S, Wei T, Gao T, Duan D, Zhao L, Li N, Li Y. The long-term effect of acupuncture for patients with chronic tension-type headache: study protocol for a randomized controlled trial. Trials. 2017 Oct 3;18(1):453. doi: 10.1186/s13063-017-2188-9. PMID 28974247